CLINICAL TRIAL: NCT04042129
Title: Urological Complications and Management After Gynecological Operations
Status: Completed | Type: Observational
Sponsor: Acibadem University (Other)
Responsible Party: Sponsor
Other Study IDs: AcibademUr
Record Dates: First submitted 2019-07-06; First posted 2019-08-01 (Actual); Last update posted 2019-08-01 (Actual); Status verified 2019-07

CONDITIONS: Urological Injury; Gynecologic Disease
MeSH Terms: conditions — Genital Diseases, Female

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: gynecologic operations with urologic complications
  Interventions: Other: gynecologic operations with urological complications

INTERVENTIONS:
Other: gynecologic operations with urological complications

SUMMARY:
OBJECTIVE: In the study, investigators aimed to evaluate the urological complications of gynecologic operations in a tertiary academic center and to evaluate the treatment methods of these complications.

METHODS: The files of all patients who underwent gynecological surgery between January 2016 and January 2019 were retrospectively reviewed. The age of patients with urological complications, American Anesthesia Society score, menopausal status, body mass index (BMI), preoperative hemoglobin level, postoperative hemoglobin level and hospitalization duration and number of previous surgeries were recorded. In addition, the patients with urological complications were evaluated in terms of the indications for surgery, type of surgery, type of urological complication and the way of treatment of the complication.

DETAILED DESCRIPTION:
In women, the anatomical localization of urinary and genital tracts is very close to each other. This proximity can lead to injuries during pelvic operations. Advances in gynecologic operation techniques and the growing experience of gynecologists may suggest a decrease in urological injuries. However, according to the literature, gynecologists face approximately 0.2% to 1% urinary tract injuries during pelvic surgeries. The increase in the number of recurrent surgeries and adverse situations encountered during the operations such as adhesions and anatomical variations factor into the persistence of urologic complications. Investigators aimed to evaluate the urological complications of gynecologic operations in a tertiary academic center and to evaluate the treatment methods of these complications.

The files of all patients who underwent gynecological surgery between January 2016 and January 2019 were retrospectively reviewed. The age of patients with urological complications, American Anesthesia Society score, menopausal status, body mass index (BMI), preoperative hemoglobin level, postoperative hemoglobin level and hospitalization duration and number of previous surgeries were recorded. In addition, the patients with urological complications were evaluated in terms of the indications for surgery, type of surgery, type of urological complication and the way of treatment of the complication.

ELIGIBILITY:
Inclusion Criteria:

-Gynecologic operations with urologic complications

Exclusion Criteria:

* Patients with incomplete data and patients who underwent obstetric operations
* patients aged under 18
* patients who were operated under emergency conditions

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — gynecologic operations
Study Population: gynecologic operations with urologic complications Patients' previous medical records, detailed physical examination findings, age, menopausal status, American Society of Anesthesiologists Classification (ASA) scores, and body mass indexes (BMI) were noted. Also, preoperative hemoglobin levels, postoperative hemoglobin levels, and hospitalization durations were recorded. In addition, indications for gynecologic surgery, sites of injury and management modalities of injury were recorded
Sampling Method: Probability Sample
Enrollment: 1754 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Number and type of Urological Complications and Management After Gynecological Operations | retrospective 3 years period

IPD SHARING:
Plan to Share IPD: No